CLINICAL TRIAL: NCT05166759
Title: Incidence and Clinical Characteristics of Pulmonary Hypertension Secondary to ARDS
Brief Title: Incidence and Clinical Characteristics of Pulmonary Hypertension Secondary to ARDS in the Highland
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Collaborators: Qinghai University (Other)
Responsible Party: Principal Investigator, Chun Pan, Chun Pan, Southeast University, China
Other Study IDs: ARDS in the highland
Record Dates: First submitted 2021-12-20; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-11

CONDITIONS: ARDS
MeSH Terms: interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Doppler ultrasound — Pulmonary artery pressure and right heart function will be assessed using Doppler ultrasound

SUMMARY:
The study is conducted in the affiliated hospital of Qinghai University .Patients in the department of Critical Care Medicine and Emergency Intensive Care Unit will be eligible for inclusion if they meet the Berlin criteria.Two researchers assess pulmonary artery pressure and right heart function of patients who are enrolled.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

18 to 80 years of age Meet the diagnostic criteria Receive invasive mechanical ventilation within 48 hours

-

Exclusion Criteria:

Patients with those disease will be excluded ： chronic obstructive pulmonary disease Pulmonary embolism Chronic heart failure Idiopathic pulmonary fibrosis Pulmonary hypertension Pregnant women will be excluded too.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is conducted in the affiliated hospital of Qinghai University .Patients in the department of Critical Care Medicine and Emergency Intensive Care Unit will be eligible for inclusion if they meet the Berlin criteria.Two researchers assess pulmonary artery pressure and right heart function of patients who are enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Pulmonary Hypertension Secondary to ARDS in the Highland | 20/11/2021-20/12/2022
ICU mortality ICU mortality | 20/11/2021-20/12/2022
  Mortality during treatment in ICU
28-days mortality rate | 20/11/2021-20/12/2022
  Mortality at 28 days of hospitalization

SECONDARY OUTCOMES:
Ventilator time | 20/11/2021-20/12/2022
  Ventilator time in ICU
Hospital length of stay | 20/11/2021-20/12/2022
  Total length of stay in hospital

OTHER OUTCOMES:
Right cardiac functionof Pulmonary Hypertension Secondary to ARDS in the Highland | 20/11/2021-20/12/2022

CONTACTS AND LOCATIONS:
Overall Officials: Chun Pan, MD, Principal Investigator — Qinghai University
Locations (1):
- Affiliated Hospital of QingHai University, Xining, Qinghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhu P, Zhu J, Tong S, She X, Qi Z, Xu Q, Shi Z, Si L, Hou M, Gan G, Pan C. Clinical characteristics of patients with a risk of pulmonary artery hypertension secondary to ARDS in a high-altitude area. BMJ Open Respir Res. 2023 Jul;10(1):e001475. doi: 10.1136/bmjresp-2022-001475. PMID 37524522